CLINICAL TRIAL: NCT06751784
Title: Randomized Placebo-controlled Phase II Cross-over Study on the Influence of Fampridine on Working Memory in Mild to Moderate Depression
Brief Title: Cross-over Study on the Influence of Fampridine on Working Memory in Mild to Moderate Depression
Acronym: FamD_2025
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christiane Gerhards, Medical Doctor, University of Basel
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2024-02355
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Working Memory; Mild to Moderate Depression
MeSH Terms: interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Experimental: Fampridin SR
  Active study medication consists of 15 tablets of fampridine SR 10 mg formulated for oral administration taken in the morning and evening 12 h apart without food. Tablets must be administered whole.
  There will be a washout period of at least 6.5 days equaling over 20 half-lives of the active substance fampridine (t½ = 6 h) between experimental and control intervention and up to 28 days depending on the individual scheduling of each subject.
  Interventions: Drug: Fampridine SR
- Other intervention (Placebo Comparator): 15 Identically looking placebo tablets consisting of widely identical additives formulated for oral administration.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fampridine SR — Active study medication consists of 15 tablets of fampridine SR 10 mg formulated for oral administration taken in the morning and evening 12 h apart without food. Tablets must be administered whole.
  Arms: Intervention
Other: Placebo — no active substance
  Arms: Other intervention

SUMMARY:
Cognitive deficits, including working memory deficits, are often present in depression and there are currently no effective pharmacological treatments targeting working memory deficits. Papassotiropoulos et al. (2024) has recently demonstrated that fampridine, a potassium channel blocker, can enhance working memory in healthy individuals with lower baseline performance, suggesting it may hold potential for addressing cognitive deficits in clinical populations. The primary aim of this study is to evaluate whether fampridine improves working memory performance in mild to moderate depression

DETAILED DESCRIPTION:
Randomized placebo-controlled phase II cross-over study on the influence of fampridine on working memory in mild to moderate depression The primary objective of this study is to evaluate if fampridine improves working memory in mild to moderate depression. It will also be assessed whether baseline working memory performance or subjective working memory deficits moderate the drug's effect.

The secondary objectives are to assess the influence of fampridine on different working memory functions, attention, cognitive flexibility, affective working memory and mood.

Intervention:Twice daily oral administration of 10 mg fampridine (Fampyra®) for 7.5 days with a wash-out period of at least 6.5 days Control intervention:Twice daily oral administration of placebo for 7.5 days Study population:Total of 38 participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Major depressive episode confirmed by the Mini-DIPS. Currently mild to moderate (MADRS: 7-30).
* Normotensive (BP: 90/60mmHg - 140/90mmHg). Sufficiently treated hypertensive subjects will be included.
* BMI: 19 - 34,9 kg/m2
* Age: 18 - 55 years
* Fluent in German
* IC as documented by signature

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to 4-aminopyridine
* Use of potassium channel blockers within the last 3 months
* Treatment with OCT 2 inhibitors and -substrates (e.g. cimetidine, propranolol)
* Treatment with antidepressants or antipsychotics within the last 3 months and throughout the study period
* Current intake of psychoactive drugs (e.g. benzodiazepines, antidepressants, neuroleptics).
* Other acute or chronic psychiatric disorder (e.g. psychosis, somatoform disorder, alcohol or drug abuse disorder)
* Cognitive impairment (MoCA score < 25)
* MADRS item 10 > 1 (suicidal tendency)
* Risk of lowered seizure threshold (due to e.g. sleep deprivation, withdrawal of alcohol after alcohol abuse, hyponatraemia)
* History of seizures
* Acute cerebrovascular condition
* Acute renal failure or severe renal insufficiency (creatinine clearance < 30 ml/min per 1.73 m2)
* Bradycardia < 50/min during clinical examination.
* History of malignant cancers
* Walking problems (e.g. due to dizziness)
* Other clinically significant concomitant disease states (e.g. hepatic dysfunction, cardiovascular disease, diabetes, asthma)
* Clinically significant laboratory or ECG abnormality that could be a safety issue in the study
* Severe somatic or neurological comorbidities
* Smoking including all nicotine containing smoking systems and devices (>10 cigarettes/units per day). Failure to withstand a test day without craving, due to regular consummation patterns.
* Pregnancy or breast feeding. Intention to become pregnant during the study participation.
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language or psychological problems of the participant
* Participation in another study with an investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
High-load working memory performance. | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  Letter n-back task which includes a 3-back task assessing working memory. The 3-back task requires participants to respond to a letter repeat with two intervening letters (for example, S-m-b-s-g…). Performance will be quantified with the d' measure controlling for false positives. Parallel versions (different sequences) are used for the four test days.

SECONDARY OUTCOMES:
Reaction time (for correct 3-back responses). | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  letter n-back task
Performance in a 0-back task (d') as a measure of attention. | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  Letter n-back task.Parallel versions (different sequences) are used for the four test days.
Adaptive verbal working memory capacity test (SPAN) backward. | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  The SPAN is a computer-based, adaptively administered test based on item response theory (Rasch model; Rasch, 1980). In the study, test form S2 (backward digit span) is used, which captures both storage capacity and executive functions (Baddeley, 2010). Adaptive administration allows for precise, efficient, and individually tailored assessment while minimizing floor and ceiling effects.
  Test scoring is based on the estimation of a continuous person parameter (θ) using weighted maximum likelihood (Warm, 1989). This parameter reflects the individual's latent working memory ability and is additionally converted into a digit span score with decimal precision, allowing for nuanced interpretation (Gignac & Weiss, 2015).
Verbal episodic memory performance measured by immediate and delayed word-list recall task. | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  In this test a list of 15 selected words will be presented to the participants with a rate of one word per two seconds and the participant should recall the words immediately in writing (immediate recall). Around 15 minutes later the participants are asked to recall the words again (short delay). Number of correct words recalled in each stage is considered as the participant's immediate and delayed recall score respectively. The four 15-words wordlists (A-D) out of the following test are used: Verbaler Lern-und Merkfähigkeitstest, VLMT
Lexical ability measured using a phonemic verbal fluency task (S-words). | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  Adapted from a subtest of the Regensburger Wortflüssigkeits-Test (RWT). In this task participants should name orally as many words as possible initiating with a special letter in one minute (e.g. Mary, Milk, Mouse, etc. for the letter M) the number of unique meaningful words will be considered as the participant's score.Different letters (B, K, P, M) are used for each test day.
Planning and Problem solving, key aspects of executive functioningwill be measured with the "Tower of London" (ToL) test. | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  In this test, participants will be tasked to rearrange colour balls to match a target arrangement in as few moves as possible. The raw score for planning ability (number of correctly solved trials with the minimum number of ball placements) is consider as the participants score. Parallel version will be used for the four test days.
Cognitive Flexibility will be assessed through the "Intra-Extra Dimensional Set Shifting (IED)" task. | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  Participants are asked to use the given feedback to work out a rule that determines which stimulus (shapes and lines in different combinations) is correct. After six correct responses, the stimuli and/or rule changes. The shifts in rule are initially intra-dimensional and then later extra-dimensional. The highest reached level is considered as the participant's score. Parallel version will be used for the four test days.
The severity of depressive symptoms will be assessed using MADRS-s (self-rating). | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  The MADRS-s consists of 9 items assessing subjects' mood, inner tension, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life. Each item is scored between 0 and 6. The total score is calculated by summing the answers of the 9 items, ranging between 0 and 54 (higher scores indicate increased severity).
The affective working memory will be assessed using an emotioanl 2-back. | Before first intake of study medication and after last intake of study medication of the 7.5-days-treatment periods
  The task follows a classic N-back paradigm with two conditions: 0-back and 2-back.
  Emotional faces (happy, sad, neutral; male/female) from the Karolinska Directed Emotional Faces set (Lundqvist et al., 1998) are presented for 1500 ms with a 1350 ms inter-stimulus interval.
  Participants indicate whether each stimulus is a "hit" or "non-hit," based on the current stimulus (0-back) or compared to the stimulus two trials prior (2-back).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, Prof. MD, Study Chair — Research Cluster Molecular and Cognitive Neurosciences; Andreas Papassotiropoulos, Prof.MD, Study Chair — Research Cluster Molecular and Cognitive Neurosciences; Annette Bruehl, Prof.MD, Study Chair — Zentrum für Affektive -, Stress- und Schlafstörungen & Zentrum für Alterspsychiatrie UPK Basel
Locations (1):
- University of Basel, Reserach Cluster Molecular and Cognitive Neurosciences, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD (de-identified) that underline results in a publication will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: PD will be available after publication, study protocol (including statistical analysis plan) will be made available before start of the study.
Access Criteria: All IPD (de-identified) that underline results in a publication will be shared upon reasonable request for scientific purposes. A reasonable request consists of a short description of the scientific purpose. Request will be reviewed by the team of the principal investigator.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: CTP FamD version 7 (2025-11-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT06751784/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: CTP FamD version 6 (2025-10-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT06751784/Prot_SAP_000.pdf